CLINICAL TRIAL: NCT04385901
Title: Long Term Functional Outcomes of COVID-19 Patients Treated by Rehabilitation Services viaTelehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Y Stone, Manager, Clinical Rehabilitative Services, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID19Recovery
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV 2; SARS Pneumonia
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients receiving care through the program developed by the University of Missouri Healthcare system will, if willing, return for follow up testing and be compared against a matched group that did not receive the rehabilitative treatment to see if there are short or long term differences.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care providers will know which group they are in, but data will be deidentified and blinded prior to analysis or viewing by the primary investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): These are patients who were diagnosed with COVID19 and recovered with usual care prior to implementation of the rehabilitation program developed by MUHC therapists. These patients will be selected in such a way as to match the approximate demographics that exist within the treatment group. These patients received education and supportive care only.
- Rehabilitation Group (Experimental): These are patients who were diagnosed with COVID19 and participated in the physical and pulmonary rehabilitation program developed at MU Healthcare as described in the study design.
  Interventions: Behavioral: Therapy Intervention

INTERVENTIONS:
Behavioral: Therapy Intervention — Patients receive 2-4 visits (based on patient presentation and need) of physical therapy, up to 4 visits of occupational therapy, up to 4 visits of speech therapy based on need. Treatment focuses on physical strengthening, pulmonary strengthening/breathing exercises, and cognitive rehabilitation.
  Arms: Rehabilitation Group

SUMMARY:
This study seeks to assess the impact of physical and pulmonary rehabilitation on patients who have been diagnosed with COVID-19 in the short and long term in hopes of establishing a best practices protocol for treatment of future patients with this disease.

DETAILED DESCRIPTION:
The novel coronavirus that began in Wuhan, China in late 2019 made an appearance in the United States in January 2020. It is a respiratory disease spreading rapidly from person to person. Recent data shows that fibrosis is seen on the lungs, and possible myocardial damage. Data shows that physical therapy was not highly utilized in recovery for these patients due to high PPE demands, and increased risk of exposure. This study will be using telehealth services to assess and treat these patients so Physical Therapy guidance is provided for movement and returning to prior level of function. Currently there is no data showing the long term effects of the those who were able to utilize Physical Therapy in recovering from COVID-19 This study will be looking at the differences in outcomes of COVID-19 positive subjects who able to complete Physical Therapy Telehealth visits versus those who did not. All groups will be tested at multiple data points for lung capacity, upper and lower extremity strength, and overall endurance to determine the long term functional effects. The control group were diagnosed with COVID-19 and recovered before the Physical and Pulmonary protocol was implemented.

ELIGIBILITY:
Inclusion Criteria:

* >Age of 18
* Positive COVID-19 diagnosis in the last 6 months

Exclusion Criteria:

* Age of <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-09-19 (Actual)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test | From 6 to 24 months post diagnosis
  Validated test demonstrating functional gait capacity and endurance; measuring change in capacity over time in 6 month increments.
Change in Short Form 35 (SF-36) Questionnaire | From 6 to 24 months post diagnosis
  Validated questionnaire assessing function and quality of life for patients with pulmonary function issues

SECONDARY OUTCOMES:
Change in Strength testing | From 6 to 24 months post diagnosis
  Use of grip dynamometer and isokinematic lower extremity testing to determine muscle capacity
Change in Peak Flow Meter Test | From 6 to 24 months post diagnosis
  Measures lung output capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Missouri Orthopedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang F, Liu N, Hu JY, Wu LL, Su GS, Zhong NS, Zheng ZG. [Pulmonary rehabilitation guidelines in the principle of 4S for patients infected with 2019 novel coronavirus (2019-nCoV)]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):180-182. doi: 10.3760/cma.j.issn.1001-0939.2020.03.007. Chinese. PMID 32164083
- [Result] Holland AE, Hill CJ, Rochford P, Fiore J, Berlowitz DJ, McDonald CF. Telerehabilitation for people with chronic obstructive pulmonary disease: feasibility of a simple, real time model of supervised exercise training. J Telemed Telecare. 2013 Jun;19(4):222-6. doi: 10.1177/1357633x13487100. Epub 2013 May 23. PMID 23666438
- [Result] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Result] Busija L, Pausenberger E, Haines TP, Haymes S, Buchbinder R, Osborne RH. Adult measures of general health and health-related quality of life: Medical Outcomes Study Short Form 36-Item (SF-36) and Short Form 12-Item (SF-12) Health Surveys, Nottingham Health Profile (NHP), Sickness Impact Profile (SIP), Medical Outcomes Study Short Form 6D (SF-6D), Health Utilities Index Mark 3 (HUI3), Quality of Well-Being Scale (QWB), and Assessment of Quality of Life (AQoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S383-412. doi: 10.1002/acr.20541. No abstract available. PMID 22588759